CLINICAL TRIAL: NCT00847236
Title: Protocol For The Quantitation Of Pain In The Diagnosis Of Polymyalgia Rheumatica
Status: Completed | Type: Observational
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-078
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Polymyalgia Rheumatica; Rheumatoid Arthritis; Rheumatic Disease
Keywords: Polymyalgia Rheumatica; Rheumatoid Arthritis; Rheumatic Disease; PMR
MeSH Terms: conditions — Polymyalgia Rheumatica; Arthritis, Rheumatoid; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Subjects with Polymyalgia Rheumatica: 50 subjects with Polymyalgia Rheumatica, both acute and chronic
- Subjects w/o Polymyalgia Rheumatica: 50 subjects with Rheumatic Disease other than polymyalgia Rheumatica
- Subjects w/o Rheumatic Disease: 50-Non Rheumatic disease subjects

SUMMARY:
The aim of this study is to evaluate a simple and rapid method in order to better define and treat Polymyalgia Rheumatica by measuring levels of muscle achiness and pain with a blood pressure cuff.

DETAILED DESCRIPTION:
This study is being conducted to evaluate a method for the quantifying of the proximal tenderness in patients with presumed diagnosis of Polymyalgia Rheumatica(PMR)using the measurements of pain thresholds(in both upper and lower arms) by the use of a standard blood pressure cuff.

At the present time the diagnosis of PMR is based upon four classic criteria, History of sudden onset symmetric painful proximal myopathy, Physical demonstrating proximal tenderness without loss of motion passively, Laboratory evidence of significant inflammation: ESR>50 and treatment with a rapidly beneficial response to low dose prednisone.

While the history, laboratory findings, and the response to prednisone are easily documented, the complaint of tenderness and the physical response to that tenderness is difficult to define and quantitate.

By better quantifying the tenderness and the physical response to that tenderness will, it is hoped, lead to more rapid diagnosis as well as improved approach to treatment.

Three groups of patients will be studied. Each patient, after written informed consent and procedure statement, will have pain threshold measurements taken and recorded by standard blood pressure cuff 4 times: one each on the lower and upper arms. The blood pressure cuff will be inflated to the level of maximum pain, then deflated, recording the maximum pain level. Absolute numbers will be used for each measurement. Blood pressure will not be recorded.

This study is an attempt to add definition to the diagnosis of Polymyalgia Rheumatica with a both simple and rapid office exam.

ELIGIBILITY:
Inclusion Criteria:

* Patients signing Informed Consent

Exclusion Criteria:

* Patients less than 50 years old

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients and Healthy volunteers from colleague referral and own practice
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To define whether the measurement of proximal arm tenderness can be used to diagnose and treat patients with Polymyalgia Rheumatica | One to two visits each subject

SECONDARY OUTCOMES:
Assessing the ease of measuring proximal arm tenderness | One to two visits each subject

CONTACTS AND LOCATIONS:
Overall Officials: Gerald S. Harris, M.D., Principal Investigator — Lahey Clinic, Inc. Arlingtion
Locations (1):
- Lahey Arlington, Arlington, Massachusetts, United States